CLINICAL TRIAL: NCT04112082
Title: Efficacy of Mobile Neurofeedback for Adult Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Myndlift Ltd. (Unknown)
Responsible Party: Principal Investigator, Dr. Tamir Epstein, Head of Unit for Adult Developmental Disorders, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6362-19-SMC
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: neurofeedback; Attention Deficit Hyperactivity Disorder (ADHD); attention; executive function; electroencephalogram (EEG); adult ADHD; wearable sensors
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Biofeedback, Psychology; Neurofeedback; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Neurofeedback Training (Experimental)
  Interventions: Behavioral: Mobile Neurofeedback
- Treatment as Usual (Active Comparator)
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Mobile Neurofeedback — Home-based neurofeedback training (downtrain theta, uptrain beta; training site: Cz) 4 times weekly for a 40 of total sessions over the ten-week training period. Session duration of 21 minutes for the first 20 sessions to 30 minutes for the last 20 sessions. Positive visual and auditory feedback when brainwaves are within the desired range.
  Other Names: neurotherapy; electroencephalogram (EEG) biofeedback; brainwave biofeedback
  Arms: Home-Based Neurofeedback Training
Other: Treatment as Usual — Treatment plan as part of regular care at the ADHD clinic, which may include pharmacological intervention, cognitive behavioral therapy (CBT), a combination of pharmacological intervention and CBT, or no intervention. Care will often include pharmacological intervention, with the specifics (e.g., type of medication, dosage) determined by psychiatrist recommendation considering such factors as response to previous interventions, participant characteristics, and practical constraints. Most pharmacological interventions will be stimulants (e.g., methylphenidate) with various release mechanisms. Each participant will receive an individualized dose titration and follow-up plan, including clinic visits as needed (generally 1-2 visits over the 10-week intervention period); interventions may be switched in accord with clinical judgment.
  Arms: Treatment as Usual

SUMMARY:
This study is an assessor-blind, parallel-group, controlled trial to evaluate the benefit of home-based training with a low-cost, mobile neurofeedback system (Myndlift) in adults with ADHD. Randomized controlled trials have shown significant benefit for neurofeedback, including persistent effects without the side effects of psychostimulants (i.e., diminished appetite, insomnia, anxiety, irritability). However, standard application requires clinic visits and significant expense, limiting training frequency and compromising potential efficacy. Additionally, extant evidence for efficacy comes almost exclusively from children and adolescents, with very few studies in adults. The present trial will measure the ability of home-based neurofeedback using a low-cost, user-friendly system to ameliorate symptomatology (e.g., enhancing attention, reducing impulsive behavior) in adults with ADHD. Participants will receive either neurofeedback or treatment as usual (TAU). Primary outcomes will be objective scores on a continuous performance task (CPT) and subjective report on a standardized adult ADHD symptoms questionnaire. Eligible participants recruited from an adult ADHD clinic will complete a baseline assessment (1.25 hours) including subjective questionnaires, computerized cognitive assessment, and resting-state EEG administered by a blinded assessor. The experimental group will train at home with a neurofeedback headset and tablet 4 times/week for ten weeks (session duration: 21-30 minutes). Neurofeedback will be provided via a conventional theta beta protocol in which participants train using gamified tasks, videos, or audio clips in a tablet-based app, and receive positive visual/auditory feedback when their brainwaves are in the desired range. The control group will follow the regular treatment plan set by the clinic (i.e., treatment as usual; TAU). Care may include pharmacological intervention, cognitive behavioral therapy (CBT), a combination of both, or no intervention. Care will often include pharmacological intervention (e.g., methylphenidate), with the specifics (e.g., type of medication, dosage) determined by psychiatrist recommendation. After completing the ten-week intervention period, all participants will return to the clinic for a follow-up assessment identical to the baseline assessment. It is hypothesized that home-based neurofeedback training will demonstrate non-inferiority to TAU as measured by improvement in subjective and objective symptoms.

ELIGIBILITY:
Inclusion Criteria:

* willingness to provide consent
* diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) of any type as ascertained by clinical interview conducted by a board-certified psychiatrist
* at the time of enrollment, not receiving treatment for symptoms of ADHD

Exclusion Criteria:

* comorbid psychotic or bipolar disorder or an active affective disorder
* medical disorder with potentially confounding psychiatric effects (either due to direct effects of the condition or medication effects)
* diagnosis of substance abuse disorder (SUD), sleep apnea, restless legs syndrome (RLS), or borderline intellectual functioning
* unable to attend in-clinic follow-up assessment
* antipsychotic agent in the three months prior to baseline assessment
* any selective serotonin reuptake inhibitor (SSRI) treatment in the four weeks prior to baseline
* other psychiatric medication in the two weeks prior to baseline that the principal investigator deems to be confounding
* experimental group only: plans to start stimulant medication during the course of the study (use of nutritional supplements including "prescription medical foods" is not exclusionary)
* neurofeedback treatment in the two years prior to baseline

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-12-22 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in Continuous Performance Task (CPT) Response Time | baseline, immediately after 10-week intervention period
  mean response time for correct responses on a computerized CPT
Change in Continuous Performance Task (CPT) Response Time Variability | baseline, immediately after 10-week intervention period
  standard deviation of response time for correct responses on a computerized CPT
Change in Self-Reported ADHD Symptoms | baseline, immediately after 10-week intervention period
  total score on the Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1)

SECONDARY OUTCOMES:
EEG Theta Amplitude | baseline, immediately after 10-week intervention period
  resting state fronto-central theta amplitude
EEG Beta Amplitude | baseline, immediately after 10-week intervention period
  resting state fronto-central beta amplitude
EEG Theta/Beta Ratio | baseline, immediately after 10-week intervention period
  resting state fronto-central theta/beta ratio
Continuous Performance Task (CPT) Accuracy | baseline, immediately after 10-week intervention period
  percent correct on a computerized CPT
Continuous Performance Task (CPT) Commission Errors | baseline, immediately after 10-week intervention period
  number of commission errors on a computerized CPT
Continuous Performance Task (CPT) Omission Errors | baseline, immediately after 10-week intervention period
  number of commission errors on a computerized CPT
ADHD Screener Score | baseline, immediately after 10-week intervention period
  sum of item scores for the first 6 items (Part A) of the Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1); item ratings: 0=never, 1=rarely, 2=sometimes, 3=often, 4=very often; scoring: for items 1-3, ratings of sometimes, often, or very often are assigned one point; for items 4-6 ratings of often or very often are assigned one point; a higher score reflects a worse outcome
ADHD Symptom Inattention Subtype Score | baseline, immediately after 10-week intervention period
  sum of item scores for the 9 inattention items from the Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1): items 1-4 & 7-11; item ratings: 0=never, 1=rarely, 2=sometimes, 3=often, 4=very often; scoring: for items 1-3 & 9, ratings of sometimes, often, or very often are assigned one point; for items 4, 7, 8, 10 & 11, ratings of often or very often are assigned one point; a higher score reflects a worse outcome
ADHD Symptom Hyperactivity/Impulsivity Subtype Score | baseline, immediately after 10-week intervention period
  sum of item scores for the 9 hyperactivity/impulsivity items from the Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1): items 5-6 & 12-18; item ratings: 0=never, 1=rarely, 2=sometimes, 3=often, 4=very often; scoring: for items 12 & 18, ratings of sometimes, often, or very often are assigned one point; for items 5-6 & 13-17, ratings of often or very often are assigned one point; a higher score reflects a worse outcome
Global Cognitive Score from Cognitive Battery | baseline, immediately after 10-week intervention period
  global cognitive score (average of standardized domain scores) from a computerized cognitive battery; scale: age- and education-adjusted mean: 100; standard deviation: 15
Attention Domain Score from Cognitive Battery | baseline, immediately after 10-week intervention period
  standardized attention domain score from a computerized cognitive battery; scale: age- and education-adjusted mean: 100; standard deviation 15
Executive Function Domain Score from Cognitive Battery | baseline, immediately after 10-week intervention period
  standardized executive function domain score from a computerized cognitive battery; scale: age- and education-adjusted mean: 100; standard deviation 15
Information Processing Speed Domain Score from Cognitive Battery | baseline, immediately after 10-week intervention period
  standardized information processing speed domain score from a computerized cognitive battery; scale: age- and education-adjusted mean: 100; standard deviation 15

OTHER OUTCOMES:
Quality of Life Scores for Adult ADHD | baseline, immediately after 10-week intervention period
  Adult ADHD Quality-of-Life Scale (AAQoL) overall score (29 items); life productivity (11 items), psychological health (6 items), life outlook (7 items), relationships (5 items) subscores from Adult ADHD Quality-of-Life Scale (AAQoL); items rated on five-point Likert scale from 'not at all/never' (1) to 'extremely/very often' (5); overall and subscale scores computed by reversing item scores for negatively worded items and transforming item scores to a 0-100 point scale; item scores summed and divided by item count; a higher score reflects a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tamir Epstein, MD, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler LA, Spencer T, Faraone SV, Kessler RC, Howes MJ, Biederman J, Secnik K. Validity of pilot Adult ADHD Self- Report Scale (ASRS) to Rate Adult ADHD symptoms. Ann Clin Psychiatry. 2006 Jul-Sep;18(3):145-8. doi: 10.1080/10401230600801077. PMID 16923651
- [Background] Brod M, Johnston J, Able S, Swindle R. Validation of the adult attention-deficit/hyperactivity disorder quality-of-life Scale (AAQoL): a disease-specific quality-of-life measure. Qual Life Res. 2006 Feb;15(1):117-29. doi: 10.1007/s11136-005-8325-z. PMID 16411036
- [Background] Schweiger A, Abramovitch A, Doniger GM, Simon ES. A clinical construct validity study of a novel computerized battery for the diagnosis of ADHD in young adults. J Clin Exp Neuropsychol. 2007 Jan;29(1):100-11. doi: 10.1080/13803390500519738. PMID 17162726
- [Background] Micoulaud-Franchi JA, Geoffroy PA, Fond G, Lopez R, Bioulac S, Philip P. EEG neurofeedback treatments in children with ADHD: an updated meta-analysis of randomized controlled trials. Front Hum Neurosci. 2014 Nov 13;8:906. doi: 10.3389/fnhum.2014.00906. eCollection 2014. PMID 25431555
- [Background] Arns M, de Ridder S, Strehl U, Breteler M, Coenen A. Efficacy of neurofeedback treatment in ADHD: the effects on inattention, impulsivity and hyperactivity: a meta-analysis. Clin EEG Neurosci. 2009 Jul;40(3):180-9. doi: 10.1177/155005940904000311. PMID 19715181
- [Background] Riesco-Matias P, Yela-Bernabe JR, Crego A, Sanchez-Zaballos E. What Do Meta-Analyses Have to Say About the Efficacy of Neurofeedback Applied to Children With ADHD? Review of Previous Meta-Analyses and a New Meta-Analysis. J Atten Disord. 2021 Feb;25(4):473-485. doi: 10.1177/1087054718821731. Epub 2019 Jan 15. PMID 30646779